CLINICAL TRIAL: NCT01006668
Title: Sevoflurane Versus Propofol for Intubation in Neonatal Intensive Care
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-13; 2009-013283-39
Record Dates: First submitted 2009-10-19; First posted 2009-11-03 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Endotracheal Intubation
Keywords: Neonates; Intensive care; Endotracheal intubation; Neonates in intensive care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Administration of sevoflurane (SEVORANE) by inhalation until a maximal concentration of 4% of inspired gas.
  Interventions: Drug: Administration of sevoflurane
- Propofol (Active Comparator): Administration of propofol (DIPRIVAN) by intravenous injection (1 mg/kg to turn over twice if necessary
  Interventions: Drug: Administration of propofol

INTERVENTIONS:
Drug: Administration of sevoflurane — Administration of sevoflurane (SEVORANE) by inhalation until a maximal concentration of 4% of inspired gas.
  Arms: Sevoflurane
Drug: Administration of propofol — Administration of propofol (DIPRIVAN) by intravenous injection (1 mg/kg to turn over twice if necessary.
  Arms: Propofol

SUMMARY:
Endotracheal intubation is a painful and stressful procedure, which is associated with acute increases of blood pressure, intracranial pressure, bradycardia and hypoxemia with high morbidity.

The aim of the study is to compare recovery time, efficacy and tolerance in a randomized controlled study, between sevoflurane and propofol for intubation in neonates in Neonatal Intensive Care Unit.

DETAILED DESCRIPTION:
Background:

Endotracheal intubation is a painful and stressful procedure, which is associated with acute increases of blood pressure, intracranial pressure, bradycardia and hypoxemia with hight morbidity.

In 2001, in France more than 50% of intubations in neonates were performed without any premedication or anesthesia.

The most frequently used anesthesias are based on benzodiazepine or opioids. Unfortunately, these treatments are responsible for respiratory and hemodynamic adverse effects. Recently, 2 new possibilities for anesthesia before intubation has been tested: propofol was better than association of morphine, succinylcholine and atropine and we shaw that inhaled sevoflurane was better than no treatment.

The aim of the present study is to compare recovery time, efficacy and tolerance in a randomized controlled study, between sevoflurane and propofol for intubation in neonates in Neonatal Intensive Care Unit.

Objectives:

The objective of this study is to compare recovery time, efficacy and tolerance in a randomized controlled study, between sevoflurane and propofol for intubation of neonates.

Methods:

Prospective, controlled, randomized, monocentric study.

Subjects:

Neonates in neonatal intensive care requiring intubation.

Evaluation criteria:

Recovery time after intubation, facilitation of procedure, tolerance of treatment (mean arterial pressure, apnea).

ELIGIBILITY:
Inclusion Criteria:

* Neonates
* Hospitalized in neonatal intensive care unit
* Needing of an endotracheal intubation

Exclusion Criteria:

* Emergency state
* Predictable difficult endotracheal intubation
* Decrease of blood pressure
* Neurological disorders
* Morphinic treatment

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2009-11; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
To compare recovery time between sevoflurane and propofol for intubation of neonates. | 18 months

SECONDARY OUTCOMES:
To compare efficacy and tolerance between sevoflurane and propofol for intubation of neonates. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice MICHEL, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France